CLINICAL TRIAL: NCT04525664
Title: Helicobacter Pylori and Chronic Dyspepsia in Eastern Uganda
Brief Title: Assessment and Management of Chronic Dyspepsia in Eastern Uganda
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jose Saenz, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201807047
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Helicobacter Pylori Infection; Dyspepsia
Keywords: helicobacter pylori; dyspepsia; prevalence
MeSH Terms: conditions — Dyspepsia | interventions — Clarithromycin; Amoxicillin; Omeprazole; Tablets

STUDY DESIGN:
Intervention Model Description: We will use the lot quality assurance sampling (LQAS) method. Households will be selected through random sampling, and each household will be asked for a list of all people over eighteen years old. Then, a person in the household will be selected using random sampling methods and be asked if they wish to participate in the study. Willing participants will provide informed consent and will be given a questionnaire to identify common symptoms of dyspepsia . All participants who complete the questionnaire will also provide a stool specimen (if willing) for fecal antigen testing. Participants who underwent Hp eradication therapy or empiric omeprazole treatment will also be given the opportunity to complete a follow-up questionnaire following completion of their treatment regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants who test positive for Helicobacter pylori (Experimental): Participants who test positive for Helicobacter pylori by fecal antigen testing will be offered treatment with triple therapy (clarithromycin 500 mg per os twice daily, amoxicillin 1 g per os twice daily, omeprazole 40 mg per os twice daily) for 14 consecutive days. Two to four weeks following the completion of treatment, participants will repeat fecal antigen testing to confirm whether they eradicated the Helicobacter pylori.
  Interventions: Drug: Clarithromycin 500mg; Drug: Amoxicillin 1000 MG; Drug: Omeprazole 40 MG
- Patients with dyspepsia and negative for Helicobacter pylori (Experimental): Participants who report chronic dyspepsia but are negative for Helicobacter pylori by fecal antigen testing will receive daily omeprazole (20 mg per os) for one month. Their symptoms will be reassessed after completion of the month treatment.
  Interventions: Drug: Omeprazole 20 MG Oral Tablet

INTERVENTIONS:
Drug: Clarithromycin 500mg — 500 mg per os twice daily for 14 consecutive days.
  Arms: Participants who test positive for Helicobacter pylori
Drug: Amoxicillin 1000 MG — 1000 mg per os twice daily for 14 consecutive days.
  Arms: Participants who test positive for Helicobacter pylori
Drug: Omeprazole 40 MG — 40 mg per os twice daily for 14 consecutive days.
  Arms: Participants who test positive for Helicobacter pylori
Drug: Omeprazole 20 MG Oral Tablet — 20 mg per os daily for 1 month; only for patients with chronic dyspepsia and who are negative for Helicobacter pylori.
  Arms: Patients with dyspepsia and negative for Helicobacter pylori

SUMMARY:
Chronic dyspepsia, or a sensation of indigestion, remains an underdiagnosed and often inappropriately managed cause of morbidity in countries with limited medical resources. A recent questionnaire of Eastern Ugandan residents identified chronic dyspepsia as the most bothersome symptom in nearly 60% of respondents, resulting in significant morbidity and work days missed. One of the most common causes for chronic dyspepsia worldwide is infection with the stomach-adapted bacterium Helicobacter pylori (Hp), the most significant risk factor for the development of stomach cancer. In developing countries, particularly in sub-Saharan Africa, the prevalence of Hp has not been accurately determined, often owing to a lack of adequate diagnostic methods. More importantly, proper diagnosis and treatment of chronic dyspepsia would limit morbidity and mortality and help decrease the likelihood of progressing to stomach cancer.

The purposes of this study are to identify the prevalence of chronic dyspepsia among residents of eastern Uganda using a questionnaire, to assess how common Hp infection is using fecal Hp antigen test kits, and to evaluate the efficacy of Hp eradication using standard Ugandan treatment guidelines. Participants who test positive for Hp infection by fecal Hp antigen testing will be offered Hp eradication treatment in the form of two antibiotics (clarithromycin, amoxicillin) and an acid-suppression medication (omeprazole), according to the current Ugandan guidelines. Patients with chronic dyspepsia who are negative for Hp (by fecal antigen testing) will be given a one-month trial of omeprazole alone, according to current American College of Gastroenterology guidelines, and their symptoms will be reassessed. At the end of the treatment regimens, participants will have the option to complete a follow-up questionnaire and provide stool samples for fecal antigen testing (if they were Hp-positive).

DETAILED DESCRIPTION:
This will be a prospective, controlled study that will be conducted in the Namutumba district. This district was selected because in a preliminary study, the prevalence of dyspeptic symptoms in this district was found to be 57%. Namutumba District has a population of slightly over 210,000 people. The prevalence of chronic dyspepsia and their associated symptoms will be determined using a questionnaire administered to all willing participants. All participants, regardless of symptoms, will also be offered fecal Hp antigen testing. Participants found to be infected with Hp will be given a 14-day course of antibiotics, per the current Ugandan standards of care, and assessed one month following completion of treatment. Participants with chronic dyspepsia who are negative for Hp will be given daily omeprazole for one month, and their symptoms will be assessed after one month.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years or older.
* All participants must provide informed consent.
* All participants receiving medications must be able to swallow pills.

Exclusion Criteria:

* A participant's inability to understand the questions or informed consent form, either in Lusoga (the regional dialect) or English (the official language of Uganda), as determined by the study team member administering the questionnaire/informed consent.
* Age less than 18 years old.
* Participants who have used any antibiotic(s) within the past 30 days.
* Participants who have used any proton pump inhibitors within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Eradication of Helicobacter pylori among Helicobacter pylori positive participants as assessed by negative fecal antigen testing at the end of the treatment regimen | 4-6 weeks.
  Participants who initially test positive for Helicobacter pylori by fecal antigen testing will receive treatment for 14 consecutive days. Two to four weeks following treatment completion, participants will repeat fecal antigen testing to confirm eradication of Helicobacter pylori. The primary outcome measure will be the percentage of participants who initially tested positive for Helicobacter pylori and were found to be negative at the end of the treatment regimen.
Number of total participants at the beginning of the study who are positive for Helicobacter pylori, as assessed by fecal antigen testing | 7 months
  The prevalence of Helicobacter pylori within the study population will be determined by conducting fecal antigen testing in participants providing informed consent.

SECONDARY OUTCOMES:
Correlation between dyspeptic symptoms from dyspepsia questionnaire and positivity for Helicobacter pylori based on fecal antigen testing | 7 months
  Based on a validated dyspepsia questionnaire, we will correlate the prevalence and severity of chronic dyspepsia with Helicobacter pylori status (determined by fecal antigen testing).
Efficacy of omeprazole for treating dyspepsia in Helicobacter pylori-negative participants. | 7 months
  We will assess the efficacy of empiric omeprazole treatment in participants with chronic dyspepsia who are negative for Helicobacter pylori by fecal antigen testing. Efficacy of treatment will be determined by a comparison of dyspepsia scores before and after treatment, as assessed by the validated dyspepsia questionnaire.

OTHER OUTCOMES:
Safety and tolerability of treatment regimen for Helicobacter pylori. | 7 months
  Participants who are provided treatment for Helicobacter pylori will meet with study coordinators 3-5 times during the treatment regimen to assess tolerability and to report any side effects or adverse reactions to the medications. Any adverse reactions will be immediately reported to the study coordinator.

CONTACTS AND LOCATIONS:
Overall Officials: Jose B Saenz, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data related to the study protocol, statistical analysis plan, and informed consent will be shared with other researchers if and when it is requested from the study's Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF